CLINICAL TRIAL: NCT00030472
Title: A Phase II Evaluation of Liposomal Doxorubicin (Doxil) in the Treatment of Persistent or Recurrent Squamous Cell Carcinoma of the Cervix
Brief Title: Liposomal Doxorubicin in Treating Patients With Persistent or Recurrent Cancer of the Cervix
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Purpose: Treatment
Other Study IDs: CDR0000069168; GOG-0127R
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2004-09

CONDITIONS: Cervical Cancer
Keywords: recurrent cervical cancer; stage IVB cervical cancer; cervical squamous cell carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms

INTERVENTIONS:
Drug: pegylated liposomal doxorubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness liposomal doxorubicin in treating patients who have persistent or recurrent cancer of the cervix.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of doxorubicin HCl liposome in patients with persistent or recurrent squamous cell carcinoma of the cervix.
* Determine the toxicity of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive doxorubicin HCl liposome IV over 1 hour on day 1. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 22-60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma (SCC) of the cervix

  * Persistent or recurrent progressive disease
* Must have failed local therapeutic measures and considered incurable
* 1 prior chemotherapeutic regimen for SCC of the cervix required

  * Initial treatment may include high-dose therapy, consolidation, or extended therapy
* Ineligible for a higher priority GOG protocol
* At least 1 unidimensionally measurable lesion

  * At least 20 mm by conventional techniques OR
  * At least 10 mm by spiral CT scan
  * Target lesion may not be within a previously irradiated field

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* GOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Platelet count at least 100,000/mm3
* Absolute neutrophil count at least 1,500/mm3

Hepatic:

* Bilirubin no greater than upper limit of normal (ULN)
* SGOT no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No congestive heart failure
* No unstable angina
* No myocardial infarction or new cardiac arrhythmia in the past 6 months

Other:

* No active infection requiring antibiotics
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* 1 prior noncytotoxic biologic regimen (e.g., monoclonal antibodies, cytokines, or small-molecule inhibitors of signal transduction) allowed for recurrent or persistent disease (provided patient has not received a noncytotoxic cytostatic regimen for recurrent or persistent disease management)
* At least 3 weeks since prior biologic or immunologic therapy for SCC of the cervix

Chemotherapy:

* See Disease Characteristics
* No prior doxorubicin or doxorubicin HCl liposome
* 1 prior noncytotoxic cytostatic regimen allowed for recurrent or persistent disease (provided patient has not received a noncytotoxic biologic regimen for recurrent or persistent disease management)
* No other prior cytotoxic chemotherapy for recurrent or persistent disease, including retreatment with initial chemotherapy regimens
* Recovered from prior chemotherapy

Endocrine therapy:

* At least 1 week since prior hormonal therapy for SCC of the cervix
* Concurrent hormone replacement therapy allowed

Radiotherapy:

* See Disease Characteristics
* Recovered from prior radiotherapy

Surgery:

* Recovered from prior surgery

Other:

* At least 3 weeks since other prior therapy for SCC of the cervix
* No prior anticancer treatment that precludes study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-12; Primary Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter G. Rose, MD, Study Chair — MetroHealth Cancer Care Center at MetroHealth Medical Center
Locations (17):
- United States (16):
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Community Hospital of Los Gatos, Los Gatos, California
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Tufts - New England Medical Center, Boston, Massachusetts
  - Cooper University Hospital, Camden, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Abington Memorial Hospital, Abington, Pennsylvania
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas M.D. Anderson CCOP Research Base, Houston, Texas
  - Fletcher Allen Health Care - Medical Center Campus, Burlington, Vermont
- Norwegian Radium Hospital, Oslo, Norway

REFERENCES:
- [Result] Rose PG, Blessing JA, Lele S, Abulafia O. Evaluation of pegylated liposomal doxorubicin (Doxil) as second-line chemotherapy of squamous cell carcinoma of the cervix: a phase II study of the Gynecologic Oncology Group. Gynecol Oncol. 2006 Aug;102(2):210-3. doi: 10.1016/j.ygyno.2005.11.048. Epub 2006 Feb 14. PMID 16478630